CLINICAL TRIAL: NCT02185677
Title: Comparison of Cognitive and Behavioral Dysexecutive Syndrome Between Parkinsonian Form and Cerebellar Form of Multiple System Atrophy and Analysis of Correlates With an Imaging Study.
Brief Title: Cognitive and Behavioral Dysexecutive Syndrome in Multiple System Atrophy
Acronym: CogAMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2013/07
Record Dates: First submitted 2014-07-01; First posted 2014-07-09 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Multiple System Atrophy
Keywords: dysexecutive syndrome; multiple system atrophy; imaging study
MeSH Terms: conditions — Multiple System Atrophy | interventions — Actigraphy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MSA-P
  Interventions: Other: Clinical evaluation; Other: neuropsychological battery test; Other: MRI; Other: Actigraphy
- MSA-C
  Interventions: Other: Clinical evaluation; Other: neuropsychological battery test; Other: MRI; Other: Actigraphy

INTERVENTIONS:
Other: Clinical evaluation
Other: neuropsychological battery test
Other: MRI
Other: Actigraphy — Actigraphy recording will be performed during 7 days after inclusion.

SUMMARY:
The main objective of the study is to compare the score to the Behavioral Dysexecutive Syndrome Inventory (BDSI) between Parkinsonian Multiple system Atrophy MSA-P patients and cerebellar Multiple System Atrophy (MSA-C) patients matched on disease duration, age (± 7 years) and sex .

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a rare neurodegenerative disorder which is characterized by a variable combination of parkinsonism, cerebellar dysfunction, autonomic failure, and additional signs. According to the consensus criteria for the diagnosis of MSA, the presence of dementia is considered an exclusion criteria. However, several studies have reported cognitive impairment in patients with MSA, dominated by a dysexecutive syndrome. Some studies have compared the cognitive profile of MSA-P patients and MSA-C but any have studied the behavioral dysexecutive syndrome in this population. In 2010, the GREFFEX has established criteria for dysexecutive syndrome and described two distinct parts: the dysexecutive syndrome and cognitive behavioral dysexecutive syndrome. Our clinical impression is that according to the type of MSA, the dysexecutive syndrome seems to be different : the MSA-P patients seem to have a cognitive dysexecutive syndrome and the MSA-C patients a behavioral dysexecutive syndrome.

We want to compare the BDSI score between MSA-P patients and MSA-C patients matched on disease duration, age and sex The specific involvement of the cerebellum in behavioral disorders could explain the behavioral differences experienced by clinicians caring for these patients but never demonstrated. The presence of these disorders could have an impact on the relationship between the patient and the caregiver. In addition, few studies have correlated with cognitive imagery data. Therefore, the exact areas involved in cognitive and behavioral MSApatients remain poorly understood.

ELIGIBILITY:
Inclusion criteria:

* Patients suffering from "probable" MSA according to clinical consensus criteria (Gilman et al, 2008),
* Age >30
* Written informed consent
* Patient covered by the national health system
* The presence of an informant
* Blood negative dosage of the hormone béta-hCG for the women old enough to procreate

Exclusion criteria:

* UMSARS IV score > 4 points
* Pregnant woman (blood positive dosage of the hormone béta-hCG) or breast feeding
* Patient under tutelage
* Patient unable to give consent
* Against indication to perform an MRI

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from MSA-P or MSA-C
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2015-06-25 (Actual); Study Completion 2015-06-26 (Actual)

PRIMARY OUTCOMES:
Behavioral Dysexecutive Syndrome Inventory scores | At inclusion (day 0)

SECONDARY OUTCOMES:
To compare the subscores of the BDSI between MSA-P patients and MSA-C patients. | At inclusion (Day 0)
To compare the cognitive tests exploring the cognitive dysexecutive syndrome between MSA-P patients and MSA-C patients. | At inclusion (Day 0)
  * Trail making Test
  * Stroop Test
  * Modfied Card Sorting Test
  * Brixton Test
  * Verbal fluency Test
  * Six Elements Test
To research correlations between scores UMSARS and cognitive and behavioral scores for MSA-P patients and MSA-C patients. | At inclusion (Day 0)
  Assessment using the Behavioral Dysexecutive Syndrome Inventory
To compare atrophied brain areas, the anatomic and functional abnormalities of neural networks between MSA-P patients and MSA-C patients. | At inclusion (Day 0)
To research correlations between imaging abnormalities and cognitive test performance in MSA patients. | At inclusion (day 0)
Actigraphy | During 7 days after inclusion
  Sleep analysis :
  Sleep / wake cycles and sleep fragmentation

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra FOUBERT-SAMIER, MD, Principal Investigator — University Hospital, Bordeaux; Rodolphe THIEBAUT, MD, PhD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France